CLINICAL TRIAL: NCT06652386
Title: Nurse-Led Telemedicine Versus In-Person Lactation Support for Breastfeeding Initiation in Mothers of Low-Birth-Weight Infants: A Non-inferiority Randomized Controlled Trial.
Brief Title: Nurse-Led Telemedicine Versus In-Person Lactation Support for Breastfeeding Initiation of Low-Birth-Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Nadia Elsharkawy, Associtae Professor, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 530-9-2024
Record Dates: First submitted 2024-10-14; First posted 2024-10-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Nurse's Role; Telemedicine; Lactation; Breastfeeding; Low Birth Weight Infants
Keywords: Nurse's Role; Telemedicine; Lactation; Breastfeeding; Low Birth Weight infants
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: * Telemedicine Group:
    * Nursing-led lactation support via secure video conferencing platforms (e.g., Zoom for Healthcare).
    * Scheduled sessions at postpartum days 1, 3, 7, and 14.
    * Additional support available upon request.
  * In-Person Group:
    * Nursing-led lactation support at the hospital bedside and during follow-up clinic visits.
    * Scheduled sessions at postpartum days 1, 3, 7, and 14.
    * Additional support available upon request.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly assigned to either the telemedicine or in-person support group using a computer-generated randomization sequence with block sizes of varying lengths to ensure allocation concealment and they are unaware of which group they have been assigned to as well as the outcome assessor is unaware
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Group (Experimental): * Nursing-led lactation support via secure video conferencing platforms (e.g., Zoom for Healthcare).
  * Scheduled sessions at postpartum days 1, 3, 7, and 14.
  * Additional support available upon request.
  Interventions: Other: Telemedicine Group
- In-Person Group (No Intervention): * Nursing-led lactation support at the hospital bedside and during follow-up clinic visits.
  * Scheduled sessions at postpartum days 1, 3, 7, and 14.

INTERVENTIONS:
Other: Telemedicine Group — * Nursing-led lactation support via secure video conferencing platforms (e.g., Zoom for Healthcare).
  * Scheduled sessions at postpartum days 1, 3, 7, and 14.
  * Additional support available upon request.
  Arms: Telemedicine Group

SUMMARY:
Breastfeeding initiation among mothers of low birth weight (LBW) infants is crucial for neonatal health but poses significant challenges. This randomized controlled trial aims to compare the effectiveness of nursing-led telemedicine lactation support versus in-person lactation support on breastfeeding initiation rates in mothers of LBW infants. The study will utilize validated tools such as the LATCH scoring system, the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), and the State-Trait Anxiety Inventory (STAI) to assess outcomes. By evaluating these two modalities, the research seeks to inform best practices for lactation support, particularly in settings where in-person care is limited.

DETAILED DESCRIPTION:
Breastfeeding offers unparalleled health benefits for infants and mothers, including optimal nutrition, immune protection, and enhanced bonding. These benefits are especially critical for low-birth-weight infants, who are at increased risk for morbidity and mortality. Despite the recognized importance, mothers of low birth weight (LBW) infants often face barriers to initiating and maintaining breastfeeding due to factors such as neonatal intensive care unit (NICU) admissions, maternal stress, and lack of specialized support.

Telemedicine in Lactation Support Telemedicine has emerged as a promising avenue for delivering healthcare services, including lactation support. It offers increased accessibility and convenience, particularly for mothers who may face challenges attending in-person consultations. While telemedicine has been successfully implemented in various healthcare domains, its effectiveness compared to traditional in-person lactation support requires further investigation, particularly among mothers of LBW infants.

Nurses play a pivotal role in providing education, emotional support, and practical assistance to breastfeeding mothers.Understanding how nursing interventions can be optimized in telemedicine versus in-person settings is essential for enhancing breastfeeding initiation.

Objectives

* To compare breastfeeding initiation rates between mothers receiving telemedicine lactation support and those receiving in-person support.
* To assess changes in breastfeeding self-efficacy using the BSES-SF.
* To evaluate maternal satisfaction with the mode of lactation support received.
* To measure maternal anxiety and stress levels using the STAI.
* To monitor infant growth parameters up to 3 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Mothers aged ≥18 years.
* Mothers of infants with a birth weight <2,500 grams.
* Mothers intend to breastfeed.
* Access to a smartphone, tablet, or computer with internet capability for the telemedicine group.

Exclusion Criteria:

* Infants with congenital anomalies affecting feeding.
* Mothers with medical conditions contraindicating breastfeeding.
* Non-English-speaking mothers (due to resource limitations).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Breastfeeding effectiveness and initiation success. | after 6 months
  Breastfeeding effectiveness assessment wil be done by using LATCH Scoring System that incldued 5 items; Each category is scored from 0 to 2, with a maximum possible score of 10. A higher score indicates better breastfeeding effectiveness, while lower scores suggest areas needing improvement. The LATCH tool helps healthcare providers to identify and support mothers who may face challenges with breastfeeding.
Maternal satisfaction levels with lactation support received | At 4 weeks postpartum
  Maternal satisfaction levels with lactation support received will be done using Maternal Breastfeeding Evaluation Scale (MBFES). It measures maternal attitudes, perceptions, and feelings about breastfeeding over time, making it valuable for evaluating the overall breastfeeding experience, especially in terms of emotional and practical aspects. The MBFES is typically divided into three main subscales:1. Infant Satisfaction/Growth, 2. Maternal Enjoyment/Role Attainment, and 3. Lifestyle and Physical Impact.
  Mothers respond to statements on a Likert scale, typically from "strongly disagree" to "strongly agree." The total score reflects the mother's overall breastfeeding experience, with higher scores indicating a more positive experience. Lower scores may point to areas where mothers might need support or guidance, such as managing discomfort or time constraints.
Breastfeeding Self-Efficacy | at baseline (after delivery) and at 4 week postpartum
  The Breastfeeding Attrition Prediction Tool (BAPT) is a psychometric instrument developed to predict a mother's likelihood of discontinuing breastfeeding. The BAPT assesses various factors influencing breastfeeding behavior and attitudes, which can predict the attrition risk.The tool is composed of four main subscales:1. Positive Breastfeeding Sentiment,2. Negative Breastfeeding Sentiment, 3. Social and Professional Support , and 4. Perceived Barriers:
  Responses are typically recorded on a Likert scale ranging from "strongly disagree" to "strongly agree." A higher score on the "Positive Breastfeeding Sentiment" subscale indicates a stronger commitment to breastfeeding, while higher scores on the other subscales (negative sentiment, barriers) may predict higher attrition risk. The overall score gives healthcare providers insight into wheth
Exclusive Breastfeeding Duration | up to 6 months postpartum
  Duration and exclusivity of breastfeeding will be followed up by Weekly phone calls to mothers up to 6 months postpartum to collect breastfeeding data.
Infant Growth Parameter - Weight | Up to 3 months postpartum
  "Infant weight will be measured in kilograms (Kg) using a baby scale at birth, 4 weeks, and 3 months postpartum. Trained nurses will perform the measurements using standardized equipment and techniques, following World Health Organization (WHO) guidelines."
Infant Growth Parameter- Length | Up to 3 months postpartum
  Length will be measured in centimeters (cm) using a measurement tape. These anthropometric measurements will be taken by trained nurses at birth, 4 weeks, and 3 months postpartum. Standardized equipment and techniques, adhering to World Health Organization (WHO) guidelines, will be employed."
Infant Growth Parameter- Head circumference | Up to 3 months postpartum
  Head circumference will be measured in centimeters (cm) using a measurement tape. These anthropometric measurements will be taken by trained nurses at birth, 4 weeks, and 3 months postpartum. Standardized equipment and techniques, adhering to World Health Organization (WHO) guidelines, will be employed."
Maternal Anxiety and Stress | at baseline (after delivery) and at 4 week postpartum
  State-Trait Anxiety Inventory (STAI) will be used to assss the level of maternal anxiety and stress. The STAI consists of 40 self-report questions, with 20 items each for state anxiety and trait anxiety. Respondents rate how they feel "right now" (state anxiety) or how they "generally" feel (trait anxiety), typically on a 4-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, Gharbia Governorate, Egypt